CLINICAL TRIAL: NCT00099138
Title: Caloric Restriction and Aging in Humans
Brief Title: CALERIE (Washington University): Comprehensive Assessment of Long-term Effects of Reducing Intake of Energy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AG0012; 3U01AG020487 (NIH)
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2006-02

CONDITIONS: Aging
Keywords: Diet; Caloric Restriction; Exercise; Energy Metabolism; Primary Aging; Secondary Aging
MeSH Terms: conditions — Motor Activity | interventions — Caloric Restriction; Exercise

INTERVENTIONS:
Behavioral: Caloric Restriction (CR)
Behavioral: Exercise

SUMMARY:
This study is one of three CALERIE trials that test the hypothesis that a reduced calorie, nutritionally sound diet increases the length of life and prevents some age-related chronic diseases such as cancer, diabetes, and cardiovascular disease. The three sites that are participating in the CALERIE trial represent a diversity of subject populations and interventional strategies.

DETAILED DESCRIPTION:
Animal studies suggest that caloric restriction (CR), or consuming fewer calories, increases life span, and also protects against some aging-related disease processes such as artherosclerosis and type II diabetes. However, it appears that simply burning more calories through physical activity does not increase life span by itself. It is not known how CR affects humans, but based on this evidence it appears that the reduced total intake and metabolism of food is the main factor, rather than increased exercise alone.

To test this, volunteers will be placed on a program of either 20% caloric restriction or 20% increase of energy expenditure by exercise, or in a control group to be instructed in healthy living. All will be evaluated on a number of potential markers of aging, on body composition, and on risk factors for artherosclerosis and diabetes.

Participation in the study will last for 12 months. The Diet group will receive individual instruction from a registered dietician. The Exercise group will be given an individualized exercise program created by a personal trainer. The Healthy Lifestyle group will be given information on how to make healthier choices; both diet and activity will be discussed. All participants will be measured every two weeks, and will keep daily food and activity logs. All will be seen by a physician and will have lab tests done before beginning the study, at 1 month, and then 3 month intervals.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 to 60
* Women must be post-menopausal
* Normal weight to moderately overweight, (Body Mass Index [BMI] between 23 - 30)
* In good health, free of major chronic diseases or conditions
* Well motivated
* Reliable

Exclusion Criteria:

* Major chronic disease or condition that would interfere with exercise or caloric restriction (such as diabetes, coronary artery disease, significant obstructive airway disease, stroke, resting blood pressure over 170 mmHg systolic and/or 100 mmHg diastolic, history or evidence of malignancy, orthopedic or musculoskeletal problems)
* Hormone replacement therapy (DHEA, estrogen, thyroid, testosterone)
* Regular exercise twice or more per week
* Smoking
* Alcoholism
* Frequent travel

Ages: 50 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48
Dates: Start 2002-03; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John O. Holloszy, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Racette SB, Weiss EP, Obert KA, Kohrt WM, Holloszy JO. Modest lifestyle intervention and glucose tolerance in obese African Americans. Obes Res. 2001 Jun;9(6):348-55. doi: 10.1038/oby.2001.45. PMID 11399781
- [Result] Fontana L, Meyer TE, Klein S, Holloszy JO. Long-term calorie restriction is highly effective in reducing the risk for atherosclerosis in humans. Proc Natl Acad Sci U S A. 2004 Apr 27;101(17):6659-63. doi: 10.1073/pnas.0308291101. Epub 2004 Apr 19. PMID 15096581
- [Derived] Racette SB, Das SK, Bhapkar M, Hadley EC, Roberts SB, Ravussin E, Pieper C, DeLany JP, Kraus WE, Rochon J, Redman LM; CALERIE Study Group. Approaches for quantifying energy intake and %calorie restriction during calorie restriction interventions in humans: the multicenter CALERIE study. Am J Physiol Endocrinol Metab. 2012 Feb 15;302(4):E441-8. doi: 10.1152/ajpendo.00290.2011. Epub 2011 Nov 29. PMID 22127229
- [Derived] Villareal DT, Fontana L, Weiss EP, Racette SB, Steger-May K, Schechtman KB, Klein S, Holloszy JO. Bone mineral density response to caloric restriction-induced weight loss or exercise-induced weight loss: a randomized controlled trial. Arch Intern Med. 2006 Dec 11-25;166(22):2502-10. doi: 10.1001/archinte.166.22.2502. PMID 17159017